CLINICAL TRIAL: NCT04966923
Title: Phenotype and Prognosis of Patients With Breast Cancer and Pathogenic Variants of TP53 (BREAST TP53)
Brief Title: Phenotype and Prognosis of Patients With Breast Cancer and Pathogenic Variants of TP53
Acronym: BREAST-TP53
Status: Completed | Type: Observational
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Sponsor
Other Study IDs: 3.0840453
Record Dates: First submitted 2021-07-08; First posted 2021-07-19 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Breast Cancer; TP53 R337H; Li-Fraumeni Syndrome; Prognosis Breast Cancer
Keywords: Breast Cancer; TP53
MeSH Terms: conditions — Breast Neoplasms; Li-Fraumeni Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — TP53 molecular analyses were initially based on the investigation of the p.R337H mutation by polymerase chain reaction/restriction fragment length polymorphism (PCR). In this method, PCR amplicons of exon 10 of the TP53 gene were digested by the Hha I restriction enzyme and then separated by agarose gel electrophoresis. This analysis can distinguish between different genotypes at the p.R337H mutation site, identifying homozygous, heterozygous and wild-type individuals for this specific mutation. Sanger sequencing of coding and splicing regions was performed in all negative cases to investigate other variants. Amplification products of exons 2-11 of TP53 Sequencing analyses were carried out on the 3130xl Genetic Analyzer. Classification of the variant pathogenicity was done according to the American College of Medical Genetics and Genomics guidelines, using VarSome or NGS germline panel. In the control group the analyses of germline painel where performed with NGS
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Breast Cancer and documented pathogenic variant TP53: Documented pathogenic or likely pathogenic variants of TP53 were identified using blood DNA colection and localized breast cancer diagnosis by histological confirmation. All patients met Revised Chompret criteria or Li Fraumeni like syndrome or family member of carrier TP53
  Interventions: Other: No intervention in this study
- Breast Cancer and no documented pathogenic variants in genetic test: Control group with localized breast cancer and no pathogenic variants documented in a genetic test
  Interventions: Other: No intervention in this study

INTERVENTIONS:
Other: No intervention in this study — Analyses of pathogenic variant TP53 and variants in genetic test

SUMMARY:
A prospective and retrospective cohort study of patients with a documented pathogenic or likely pathogenic variants of TP53 were identified using blood DNA colection and breast cancer diagnosis by histological confirmation, between 1999 and 2022. All patients were followed by the Hereditary Group of a single cancer center (Instituto do Cancer do Estado de Sao Paulo). Patients were included if they had a histopathological diagnosis of localized invasive carcinoma or in situ carcinoma of the breast and with localized disease. Patients met Revised Chompret criteria, Li Fraumeni like syndrome,family member of carrier TP53 or hereditary breast and ovarian syndrome for germline test.

DETAILED DESCRIPTION:
The primary outcome was progression free survival from specific breast cancer from patients with BC and TP53 mutation versus BC and no pathogenic variants documented in genetic test. We proposed 45 cases TP53 pathogenic carriers and localized breast cancer diagnosed for each case included we will be selected 2 controls resulting in 90 control patients, for control with no documented pathogenic variants in genetic test. With a sample of 135 patients with distribution 2:1, considering a two-tailed alpha of 5%, the study will have 80% power to identify a hazard hatio of 0.62 in the comparison of progression-free survival between the groups.

Descriptive statistics will be used to summarize clinical characteristics and treatments performed. Continuous variables may be compared between groups using T Student test or Mann-Whitney test, in the case of normal and non-normal data distribution, respectively. Categorical variables may be compared between groups using the Fisher exact test.

Progression-free survival will be estimated from the date of breast cancer diagnosis until the date of progression or date of recurrence (in cases of localized disease treated) of breast cancer. Death will not be considered as an event for progression-free survival, since patients with PV TP53 may have an increased risk of deaths from other neoplasms. The breast cancer specific survival will be estimated from the date of diagnosis of breast cancer until the date of death from the breast cancer. Patients without the specific events will be censored on the date of last follow-up.

The Kaplan-Meyer method will be used for survival estimates, comparing survival curves with log-rank testing. The Cox regression model will be used for hazard-ratio calculation and 95% confidence-interval. P value less than 0.05 will be considered statistically significant. Statistical analyses will be performed through Stata program, version 15.1 (StataCorp, Texas, USA).

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer (histopathological diagnosis of localized invasive carcinoma or in situ carcinoma of the breast) and documented germline pathogenic variants of TP53.

Exclusion Criteria:

* Patients with only other types of breast cancer such as sarcoma and phyllodes tumor were excluded from the analysis.

  * Metastatic Breast Cancer at diagnosis ("denovo")

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A prospective and retrospective cohort study of patients with a documented pathogenic or likely pathogenic variants of TP53 were identified using blood DNA colection and breast cancer diagnosis by histological confirmation, between 1999 and 2022. All patients were followed by the Hereditary Group of a single cancer center (Instituto do Cancer do Estado de Sao Paulo). Patients were included if they had a histopathological diagnosis of localized invasive carcinoma or in situ carcinoma of the breast. All patients met Revised Chompret criteria or Li Fraumeni like syndrome or family member of carrier TP53 or hereditary breast and ovarian Syndrome. Patients with only other types of breast cancer such as sarcoma and phyllodes tumor were excluded from the analysis.
Sampling Method: Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2018-12-02 (Actual); Primary Completion 2021-08-07 (Actual); Study Completion 2022-02-22 (Actual)

PRIMARY OUTCOMES:
Progression free survival | We proposed 45 cases TP53 pathogenic carriers and breast cancer diagnosed for each case included we will be selected 2 controls resulting in 90 control patients, for control are estimated with the same age (range 10 years)
  progression free survival from specific breast cancer from patients with BC and TP53. mutation versus BC and no pathogenic variants documented in genetic test. gnosed for each case included we will be selected 2 controls resulting in 90 control patients, for control are estimated with the same age (range 10 years), staging and immunohistochemistry

SECONDARY OUTCOMES:
Overall Survival, causes of deaths, local breast cancer recurrence and contra-lateral breast cancer recurrence | This study will enrollment 45 cases TP53 pathogenic carriers and breast cancer diagnosed for each case included we will be selected 2 controls resulting in 90 control patients, for control are estimated with the same age (range 10 years)

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Petry, MD, Principal Investigator — Instituto do Cancer do Estado de São Paulo
Locations (1):
- ICESP, São Paulo, Brazil